CLINICAL TRIAL: NCT03164655
Title: A Randomized Phase II Study Comparing Treatment Intensification With CIAH Plus Systemic Chemotherapy to Systemic Chemotherapy Alone in Patients With Liver-only Colorectal Metastases Considered Still Non Resectable After at Least Two Months of Systemic Induction Chemotherapy
Brief Title: Improving SUrgery of Liver Metastases: a Trial of the Arterial Chemotherapy Network
Acronym: SULTAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCGI 30 - PRODIGE 53 SULTAN; 2016-001493-15 (EudraCT Number)
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Oxaliplatin; Cetuximab; Bevacizumab; Panitumumab; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAI oxaliplatin combined with I.V. FOLFIRI + target therapy (Experimental): * HAI oxaliplatin 100 mg/m² on D1
  * I.V. cetuximab 500 mg/m² or panitumumab 6 mg/kg or bevacizumab 5 mg/kg D1 according to RAS status and prior response/tolerance to systemic induction CT
  * modified FOLFIRI regimen without fluorouracil bolus
  * I.V. irinotecan 180 mg/m² D1
  * I.V. bolus 5-Fluorouracil (5-FU): 0
  * I.V. leucovorin 400 mg/m² in 2 hours D1
  * I.V. continuous infusion 5-FU 2400 mg/m² in 46 hours
  Interventions: Drug: Oxaliplatin, Cetuximab, Bevacizumab, Panitumumab, Irinotecan, Leucovorin, 5-Fluorouracil
- conventional systemic CT (Active Comparator): * Response to systemic induction CT
  * Toxicity and duration of the systemic induction CT
  * RAS status
  * Current guidelines/standard of care
  Interventions: Drug: Oxaliplatin, Cetuximab, Bevacizumab, Panitumumab, Irinotecan, Leucovorin, 5-Fluorouracil

INTERVENTIONS:
Drug: Oxaliplatin, Cetuximab, Bevacizumab, Panitumumab, Irinotecan, Leucovorin, 5-Fluorouracil — Oxaliplatin 100 mg/m² infusion in 2 hours, Cetuximab 500mg/m² infusion in 2 hours, Bevacizumab 5 mg/kg infusion in 30 minutes, Panitumumab 6 mg/kg, Irinotecan 180 mg/m² over 90 minutes to begin 30 minutes after folinic acid infusion is started, Leucovorin 400 mg/m² infusion in 2 hours, 5-Fluorouracil 2400 mg/m² infusion continuous in 46h

SUMMARY:
National trial, multicenter, randomized, phase II comparing treatment intensification with hepatic arterial infusion chemotherapy plus systemic chemotherapy (CT) to systemic chemotherapy alone in patients with liver-only colorectal metastases (CRLM) considered still non resectable after at least two months of systemic induction chemotherapy.

DETAILED DESCRIPTION:
to compare the efficacy of CT intensification combining hepatic arterial infusion(HAI) oxaliplatin plus IV FOLFIRI plus targeted therapy (anti-epidermal growth factor receptor (EGFR) or bevacizumab) to conventional systemic CT alone plus targeted therapy (anti-EGFR or antiangiogenic antibody), in patients with liver-only CRLM not amenable to curative-intent resection (and/or ablation) after systemic induction CT in terms of conversion to complete (R0 R1) resection (or ablation) rate (CRR).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal cancer (CRC), and radiologic or histologic proof of CRLM not amenable to a curative intent-treatment.
2. At least two months of prior induction systemic CT with oxaliplatin and/or irinotecan combined with a fluoropyrimidine combined or not to a targeted therapy (e.g., anti-EGFR or antiangiogenic antibody) for metastatic disease (patients ending their adjuvant chemotherapy after primary tumor resection since more than 6 months should also have received first-line chemotherapy for metastatic disease). Further systemic chemotherapy lines are allowed.
3. Unresectability of the CRLM will be confirmed by a centralized multidisciplinary expert panel (composed of surgeons, radiologists, interventional radiologists and medical oncologists). The panel will review the CT scan and MRI of the patients (weekly web conference). Non-resectability criteria (one of the following criteria):

   * Upfront R0/R1 resection of all CRLM (that leaves at least two adequately perfused and drained segments) is not possible
   * and/or metastases in contact with major vessels of the remnant liver which would require resection of the vessel for an R0 resection (i.e., tumor involvement of main portal right and left portal veins, of the three main hepatic veins, or of the retrohepatic vena cava)
   * and/or documented progressive disease on imaging (according to the RECIST v1.1) or doubling of serum levels of carcinoembryonic antigen (CEA) or carbohydrate antigen 19-9 (CA 19-9) following ≥2 months of induction CT
4. At least one measurable liver metastasis according to the RECIST v1.1
5. Age ≥18 years
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
7. Normal liver function, i.e. bilirubin <1.5 times the upper limit of normal values (ULN), aminotransferases <5 ULN, alkaline phosphatase <5 ULN
8. International normalized ratio (INR) <1.5 ULN
9. Neutrophils >1500/mm³, platelets >100 000/mm³, hemoglobin >9 g/dL (transfusion allowed)
10. Calculated creatinine clearance >50 mL/min (Cockcroft and Gault formula)
11. Informed consent signed by the patient or his/her legal representative
12. Patient affiliated to a social security regimen
13. Potentially reproductive patients must agree to use an effective contraceptive method or practice adequate methods of birth control or practice complete abstinence while on treatment, and for at least 6 months after the last dose of study drug.
14. Uracilemia <16 ng/ml

Exclusion Criteria:

1. Patient eligible for curative-intent treatment of CRLM (i.e. resection and/or thermoablation), according to the local multidisciplinary team and/or the central review.
2. Definitive anatomical contraindication to complete surgical resection (any of the following criteria):

   * More than two lesions in all liver segments
   * Bilobar liver metastasis and more than three lesions >3 cm in the hepatic lobe the least affected (i.e. the future remnant liver)
   * Bilobar liver metastasis and disease liver extend >50%
3. Extrahepatic tumor disease (except ≤3 lung nodules <10 mm deemed amenable to curative-intent resection/thermoablation and non-resected primary tumor with no or mild symptoms)
4. Patient with contraindication for trial drugs (investigators have to refer to drugs SmPC); contraindication limited to targeted therapy (e.g., anti-EGFR or antiangiogenic antibody) is not an exclusion criteria
5. Disease progression after FOLFOXIRI/FOLFIRINOX
6. Sensory neuropathy ≥ grade 2 (National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.4.0)
7. If patients received bevacizumab, following non-inclusion criteria must be respected:

   * Proteinuria >1 g,
   * Gastro-intestinal fistulae or perforation,
   * Hypersensitivity to Chinese hamster ovary cell products or other human recombinant antibody,
   * Major surgery in the last 28 days.
8. If patients received panitumumab, following non-inclusion criteria must be respected:

   * Interstitial lung disease,
   * Pulmonary fibrosis.
9. Significant chronic liver disease (resulting in portal hypertension and/or liver insufficiency)
10. Allergy to contrast media that cannot be managed with standard care
11. Previous organ transplantation, HIV or other immunodeficiency syndromes
12. Concomitant or past history of cancer within 5 years prior to entry into the trial other than adequately treated basal-cell skin cancer or in situ carcinoma of the cervix
13. Patients with clinically significant active heart disease or myocardial infarction in the last 6 months
14. Concomitant medications/comorbidities that may prevent the patient from receiving study treatments as uncontrolled intercurrent illness (for instance: active infection, active inflammatory disorders, inflammatory bowel disease, intestinal obstruction, uncontrolled hypertension systolic >15 and diastolic >9, symptomatic congestive heart failure…)
15. Ionic disorders as:

    * Kalemia ≥1 x ULN
    * Magnesemia <0.5 mmol/L
    * Calcemia <2 mmol/L
16. Patient with a dihydropyrimidine dehydrogenase (DPD) deficiency; Uracilemia ≥16 ng/ml, the test should be done for all patients before first 5-FU administration, according to "agence nationale de sécurité du médicament" (ANSM) communication regarding recommendation about high risk of no testing DPD in patient before 5-FU administration
17. QT/QTc >450 msec for men and > 470 msec for women
18. Concomitant intake of St. John's wort
19. Patient already included in another clinical trial with an experimental treatment
20. Pregnancy or lactation
21. Patients deprived of liberty or under guardianship
22. Patients unable to undergo medical monitoring test for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Curative-intent (R0-R1) resection (and/or ablation) rate (CRR) of CRLM | 6 months
  Curative-intent (R0-R1) resection (and/or ablation) rate (CRR) of CRLM confirmed by a systematic review of the surgical and pathological report by an independent committee blind to the treatment received

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Boige, Principal Investigator — Gustave Roussy Villejuif
Locations (4):
- France (4):
  - Ico Paul Papin, Angers
  - Centre Eugene Marquis, Rennes
  - Chp Saint Gregoire, Saint-Grégoire
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.
Access Criteria: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.

REFERENCES:
- [Derived] Boileve A, Audemar F, Dupont-Bierre E, Le Sourd S, Ulusakarya A, Chauvenet M, Benmaziame A, Wagner M, Goere D, Dromain C, Gelli M, Pezzella V, Bonnet B, Tanguy ML, Boige V. Treatment Intensification with Hepatic Arterial Infusion Chemotherapy in Patients with Liver-Only Colorectal Metastases Still Unresectable After Systemic Induction Chemotherapy: Exploratory Findings From a Prematurely Closed Multicenter Randomized Phase II Study: SULTAN UCGI 30/PRODIGE 53 (NCT03164655). Ann Surg Oncol. 2026 Feb;33(2):1460-1469. doi: 10.1245/s10434-025-18570-5. Epub 2025 Oct 21. PMID 41118066
- [Derived] Boileve A, Maillard A, Wagner M, Dromain C, Laurent C, Dupont Bierre E, Le Sourd S, Audemar F, Ulusakarya A, Guerin-Meyer V, Smisth D, Pezzella V, De Baere T, Goere D, Gelli M, Taieb J, Boige V. Treatment intensification with hepatic arterial infusion chemotherapy in patients with liver-only colorectal metastases still unresectable after systemic induction chemotherapy - a randomized phase II study -- SULTAN UCGI 30/PRODIGE 53 (NCT03164655)- study protocol. BMC Cancer. 2020 Jan 30;20(1):74. doi: 10.1186/s12885-020-6571-7. PMID 32000724